CLINICAL TRIAL: NCT00380380
Title: A Randomized, Single-blind, Placebo Controlled, Cross-over Study to Evaluate the Acute Effects of Vildagliptin on Gastric Emptying in Patients With Type 2 Diabetes.
Brief Title: A Study to Assess the Acute Effects of Vildagliptin on Gastric Emptying in Patients With Type 2 Diabetes.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CLAF237A2378
Record Dates: First submitted 2006-09-22; First posted 2006-09-26 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Vildagliptin, type 2 diabetes, gastric emptying
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin

SUMMARY:
Please note this study is not being conducted in the United States. The purpose of this study is to assess the acute effects of vildagliptin, an unapproved drug, in reducing post-meal glucose levels by delaying gastric emptying.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to complete a 1-week wash-out of current anti-diabetic medications
* Cannot take any medications which may alter gastric motility except for cardiac medication at a stable dose
* Blood glucose criteria must be met
* BMI <40

Exclusion Criteria:

* History of type 1 diabetes, diabetes resulting from pancreatic injury, or secondary forms of diabetes
* Need for insulin within 3 months or patients on thiazolidinediones
* Significant concommitant disease or complications of diabetes
* Patients with any history of gastrointestinal surgery or positive gastrointestinal symptons
* Abnormal liver function tests as defined by the protocol
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 30 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2006-01; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the effects of acute effects of vildagliptin on gastric emptying

SECONDARY OUTCOMES:
Effect on steady state levels of active GLP-1 and GIP
Change in fasting and postprandial glucose levels.
Change in glucagon secretion
Change in postprandial glucose kinetics
Effect on gastric peristalsis
Effect on satiety

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Munich, 81377, Germany, Munich, Germany

REFERENCES:
- [Result] Vella A, Bock G, Giesler PD, Burton DB, Serra DB, Saylan ML, Dunning BE, Foley JE, Rizza RA, Camilleri M. Effects of dipeptidyl peptidase-4 inhibition on gastrointestinal function, meal appearance, and glucose metabolism in type 2 diabetes. Diabetes. 2007 May;56(5):1475-80. doi: 10.2337/db07-0136. Epub 2007 Feb 15. PMID 17303799